CLINICAL TRIAL: NCT05648071
Title: Sintilimab Plus Bevacizumab and Platinum-Based Doublet Chemotherapy as First-Line Treatment for Advanced Non-squamous Non-Small-Cell Lung Cancer With Negative Driver Gene: a Single-center, Single-Arm Trial
Brief Title: First-Line Treatment for Advanced Non-squamous Non-Small-Cell Lung Cancer With Negative Driver Gene: a Single-center, Single-Arm Trial
Acronym: SPBPDC
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Qianfoshan Hospital (Other)
Responsible Party: Principal Investigator, Degan Lu, professor, Qianfoshan Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YXLL-KY-2022(036)
Record Dates: First submitted 2022-12-04; First posted 2022-12-13 (Actual); Last update posted 2022-12-13 (Actual); Status verified 2022-12

CONDITIONS: Advanced Non-squamous Non-Small-Cell Lung Cancer
Keywords: Non-squamous Non-Small-Cell Lung Cancer,Sintilimab, Bevacizumab
MeSH Terms: interventions — sintilimab; Bevacizumab; Pemetrexed; nedaplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sintilimab Plus Bevacizumab and Platinum-Based Doublet Chemotherapy (Experimental): The specific treatment regimen is as follows :Non-squamous NSCLC: Sintilimab (200 mg) plus Bevacizumab (7.5mg/kg) is started on the first day of each treatment cycle and administered every three weeks. Nedaplatin (80-100 mg/m2) (d2) +pemetrexed 500 mg/m2 (d2) Q3W is administered in this regimen for 4 cycles followed by sintilimab plus bevacizumab until disease progression or intolerable toxicity.
  Interventions: Drug: Sintilimab

INTERVENTIONS:
Drug: Sintilimab — The specific treatment regimen is as follows :Non-squamous NSCLC: Sintilimab (200 mg) plus Bevacizumab (7.5mg/kg) is started on the first day of each treatment cycle and administered every three weeks. Nedaplatin (80-100 mg/m2) (d2) +pemetrexed 500 mg/m2 (d2) Q3W is administered in this regimen for 4 cycles followed by sintilimab plus Bevacizumab until disease progression or intolerable toxicity.
  Other Names: Bevacizumab; Pemetrexed; Nedaplatin

SUMMARY:
To evaluate the efficacy and safety of sintilimab plus bevacizumab and platinum-based doublet chemotherapy as the first-line therapy for advanced nonsquamous non-small-cell lung cancer(NSCLC) with negative driver gene.

This study is an exploratory single-arm study. The specific treatment regimen is as follows: Non-squamous NSCLC: Sintilimab (200 mg) plus Bevacizumab (7.5mg/kg) is started on the first day of each treatment cycle and administered every three weeks. Nedaplatin (80-100 mg/m2) (d2) +pemetrexed 500 mg/m2 (d2) Q3W is administered in this regimen for 4 cycles followed by sintilimab plus bevacizumab until disease progression or intolerable toxicity.

Patients are assessed for measurable disease at baseline, 6 weeks, 12 weeks after starting treatment, and every 9 weeks thereafter according to RECIST 1.1 criteria during the treatment period until disease progression or intolerable toxicity withdrawal. Following discontinuation of treatment, subjects are followed for survival status every 3 months until death. Subject safety was assessed during treatment according to NCI CTCAE Version 4.0 criteria. Subjects who experience an AE should be followed until the AE returns to baseline. The primary endpoints is Progression-free survival (PFS) . Secondary endpoints include objective response rate (ORR), overall survival (OS) and safety (NCI CTCAE v 4.0). Statistical methods: The PFS curve was estimated using the Kaplan-Meier method for the largest population to be analyzed. The confidence interval method was used as the criterion for the main analysis. OS was calculated in the same way as the secondary endpoint. Descriptive statistics will be used to analyze ORR, DCR, etc. It is expected that sintilimab plus bevacizumab and platinum-based doublet chemotherapy as first-line treatment will prolong median PFS and OS in patients with driver gene-negative advanced Non-squamous NSCLC.

DETAILED DESCRIPTION:
Lung cancer is the most common cause of cancer mortality worldwide[1]. NSCLC represents more than 80% of lung cancer cases[2], with most having nonsquamous histology[3].Current first-line treatment options in metastatic nonsquamous NSCLC without oncogenic driver alterations include checkpoint inhibitor monotherapy in patients with high programmed death-ligand 1 (PD-L1) expression and checkpoint inhibitor therapy in combination with platinum-doublet chemotherapy with or without bevacizumab[4.5].Despite the available standard-of-care first-line treatments, clinical outcomes have remained suboptimal and additional therapeutic options are needed.

Sintilimab is a recombinant, fully human IgG4 anti-PD-1 monoclonal antibody. Preclinical data have shown that sintilimab has a greater affinity against PD-1 than pembrolizumab or nivolumab[6].In a randomised, double-blind, phase 3 trial, sintilimab plus chemotherapy resulted in significantly longer progression-free survival and overall survival versus chemotherapy alone in patients with treatment-naive NSCLC without EGFR or ALK genomic tumour mutations, with a manageable safety profile[7.8].

Bevacizumab, in addition to its known anti-angiogenic effects, has immunomodulatory effects through inhibition of vascular endothelial growth factor (VEGF), including promotion of dendritic cell maturation; normalisation of the tumour vasculature, which might increase T-cell infiltration; and reprogramming of the tumour microenvironment from being immune suppressive to immune permissive[9.10]. Therefore, reversal of VEGF-mediated immunosuppression by bevacizumab could enhance the antitumour activity of sintilimab.

We aimed to evaluate the efficacy and safety of sintilimab with bevacizumab plus platinum-based doublet chemotherapy for the treatment of patients with driver gene-negative advanced nonsquamous NSCLC.

Objective: To evaluate the efficacy and safety of sintilimab plus bevacizumab and platinum-based doublet chemotherapy as the first-line therapy for advanced nonsquamous non-small-cell lung cancer with negative driver gene.

The research idea starts from the safety and efficacy of sintilimab plus bevacizumab and platinum-based doublet chemotherapy for NSCLC. Under the theoretical perspective of clinical research on cancer treatment, an exploratory single-center single-arm study method is used to perform sintilimab plus bevacizumab and platinum-based doublet chemotherapy regimen for first-line treatment of advanced nonsquamous NSCLC patients with negative driver gene. A database is established for the enrolled case report form, systematic data analysis is performed, and finally the study conclusions of above treatment safety and efficacy are obtained. It is expected that sintilimab plus bevacizumab and platinum-based doublet chemotherapy as first-line treatment will prolong median PFS and OS in patients with driver gene-negative advanced nonsquamous NSCLC.

This study is an exploratory single-arm study. The specific treatment regimen is as follows :Non-squamous NSCLC: Sintilimab (200 mg) plus Bevacizumab (7.5mg/kg) is started on the first day of each treatment cycle and administered every three weeks. Nedaplatin (80-100 mg/m2) (d2) +pemetrexed 500 mg/m2 (d2) Q3W is administered in this regimen for 4 cycles followed by sintilimab plus Bevacizumab until disease progression or intolerable toxicity.

Patients are assessed for measurable disease at baseline, 6 weeks, 12 weeks after starting treatment, and every 9 weeks thereafter according to RECIST1.1 criteria during the treatment period until disease progression or intolerable toxicity withdrawal. Following discontinuation of treatment, subjects are followed for survival status every 3 months until death. Subject safety was assessed during treatment according to NCI CTCAE Version 4.0 criteria. Subjects who experience an AE should be followed until the AE returns to baseline. The primary endpoints is Progression-free survival (PFS) . Secondary endpoints include objective response rate (ORR), overall survival (OS) and safety (NCI CTCAE v 4.0).

Statistical methods: The PFS curve was estimated using the Kaplan-Meier method for the largest population to be analyzed. The confidence interval method was used as the criterion for the main analysis. OS was calculated in the same way as the secondary endpoint. Descriptive statistics will be used to analyze ORR, DCR, etc.

ELIGIBILITY:
Inclusion Criteria:

1. Metastatic Non-squamous NSCLC is histologically or cytologically proven to be inoperable and cannot receive radical concurrent chemoradiotherapy. The conventional TNM stage was identified as stage IIIa-Ⅳb according to the International Association for the Study of Lung Cancer and the American Joint Committee on the Classification of Cancer 8th edition TNM Staging of Lung Cancer.
2. Patients with driver-negative advanced Non-squamous NSCLC.
3. Patients who had not previously received systemic radiotherapy and chemotherapy or who had relapsed for more than 6 months of follow-up after onset of adjuvant chemotherapy.
4. At least one measurable lesion as determined by RECIST criteria.
5. Male or female patients, age: 18-75 years of age.
6. Performance score 0-1 based on Eastern Cooperative Oncology Group (ECOG) test.
7. Expected survival period ≥12 weeks.
8. Serum absolute number of neutrophils≥ 1.5 x 10^9/L, platelet ≥ 100 x10^9/L, and hemoglobin≥ 90g/L.
9. Serum bilirubin≤1.5 times ULNL, aspartate aminotransferase (AST) and adenosine triphosphate(ALT) ≤ 2.5 times ULN, alkaline phosphatase ≤ 5 times ULN.
10. Serum creatinine≤ the ULN or creatinine clearance ≥ 60 mL/min.
11. Patients who had previously undergone surgery have recovered for more than 4 weeks from the beginning of the project.
12. Women with an intact uterus must have a negative pregnancy test within 28 days prior to enrolement in the study (unless it was 24 months after amenorrhea). If the pregnancy test is more than 7 days prior to initial dosing, a urine pregnancy test is required for verification (within 7 days prior to initial dosing).
13. If there is a risk of conception, all patients (whether male or female) are required to use contraceptive measures with an annual failure rate of less than 1% throughout the treatment period until 120 days after the last dose of the study drug.
14. Sign the inform consent form with good compliance.

Exclusion criteria:

1. Those who are known to be allergic to the study drug sintilimab, bevacizumab and and its any components.
2. Intolerance to study drug treatment or allergy to the active ingredients or excipients of combined chemotherapy drugs.
3. Pregnancy or breastfeeding women or women who may be pregnant but are unwilling to take appropriate contraception.
4. Existing severe acute infections that are not under control; Or suppurative and chronic infections with delayed healing.
5. Pre-existing serious heart disease, including: congestive heart failure, uncontrolled high-risk arrhythmias, unstable angina pectoris, myocardial infarction, severe valvular heart disease, and refractory hypertension.
6. People suffering from uncontrollable neuropsychiatric diseases or mental disorders had poor compliance and were unable to cooperate and describe treatment responses; The conditions of patients with primary brain tumor or central nerve metastatic tumor were uncontrollable and the symptoms of cranial hypertension or neuropsychiatric were obvious.
7. Patients with hereditary bleeding tendency or coagulation dysfunction, or history of thrombosis or bleeding, and abnormal detection results of coagulation function related indicators.
8. Patients who are receiving thrombolytic or anticoagulant therapy due to high risk of thrombosis.
9. Patients with unhealed wounds, unhealed ulcers or unhealed fractures.
10. Other conditions that the investigator considers to be inappropriate for the patient to participate in this trial.
11. Currently participating in interventional clinical research treatment, or have received other investigational drugs or used investigational device treatment within 4 weeks before the first dose.
12. Patients who have undergone major surgery within 4 weeks before the start of study treatment or are scheduled to undergo major surgery during the study period (except for surgery such as puncture or lymph node biopsy).
13. Pulmonary interstitial fibrosis with respiratory failure.
14. Chronic obstructive pulmonary disease with respiratory failure.
15. Active pulmonary tuberculosis;
16. Active autoimmune disease requiring systemic therapy (such as the use of disease-modifying drugs, glucocorticoids, or immunosuppressants) within 2 years prior to the first dose. Replacement therapy (such as thyroxine) is not considered systemic therapy;
17. Those who are receiving systemic glucocorticoid therapy (excluding nasal spray, inhalation or other local glucocorticoids) or any other form of immunosuppressive therapy within 14 days before the first dose of the study;
18. Have previously received the following therapies: anti-pd1 drugs, anti-PD-L1 drugs.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
PFS | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 36 months
  Progression-free survival

SECONDARY OUTCOMES:
OS | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 36 months
  overall survival
ORR | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 36 months
  objective response rate
DOR | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 36 months
  Duration of Responst

CONTACTS AND LOCATIONS:
Overall Officials: Degan Lu, professor, Principal Investigator — Shandong First Medical University
Locations (1):
- The First Affiliated Hospital of Shandong First Medical University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Global Burden of Disease Cancer Collaboration; Fitzmaurice C, Abate D, Abbasi N, Abbastabar H, Abd-Allah F, Abdel-Rahman O, Abdelalim A, Abdoli A, Abdollahpour I, Abdulle ASM, Abebe ND, Abraha HN, Abu-Raddad LJ, Abualhasan A, Adedeji IA, Advani SM, Afarideh M, Afshari M, Aghaali M, Agius D, Agrawal S, Ahmadi A, Ahmadian E, Ahmadpour E, Ahmed MB, Akbari ME, Akinyemiju T, Al-Aly Z, AlAbdulKader AM, Alahdab F, Alam T, Alamene GM, Alemnew BTT, Alene KA, Alinia C, Alipour V, Aljunid SM, Bakeshei FA, Almadi MAH, Almasi-Hashiani A, Alsharif U, Alsowaidi S, Alvis-Guzman N, Amini E, Amini S, Amoako YA, Anbari Z, Anber NH, Andrei CL, Anjomshoa M, Ansari F, Ansariadi A, Appiah SCY, Arab-Zozani M, Arabloo J, Arefi Z, Aremu O, Areri HA, Artaman A, Asayesh H, Asfaw ET, Ashagre AF, Assadi R, Ataeinia B, Atalay HT, Ataro Z, Atique S, Ausloos M, Avila-Burgos L, Avokpaho EFGA, Awasthi A, Awoke N, Ayala Quintanilla BP, Ayanore MA, Ayele HT, Babaee E, Bacha U, Badawi A, Bagherzadeh M, Bagli E, Balakrishnan S, Balouchi A, Barnighausen TW, Battista RJ, Behzadifar M, Behzadifar M, Bekele BB, Belay YB, Belayneh YM, Berfield KKS, Berhane A, Bernabe E, Beuran M, Bhakta N, Bhattacharyya K, Biadgo B, Bijani A, Bin Sayeed MS, Birungi C, Bisignano C, Bitew H, Bjorge T, Bleyer A, Bogale KA, Bojia HA, Borzi AM, Bosetti C, Bou-Orm IR, Brenner H, Brewer JD, Briko AN, Briko NI, Bustamante-Teixeira MT, Butt ZA, Carreras G, Carrero JJ, Carvalho F, Castro C, Castro F, Catala-Lopez F, Cerin E, Chaiah Y, Chanie WF, Chattu VK, Chaturvedi P, Chauhan NS, Chehrazi M, Chiang PP, Chichiabellu TY, Chido-Amajuoyi OG, Chimed-Ochir O, Choi JJ, Christopher DJ, Chu DT, Constantin MM, Costa VM, Crocetti E, Crowe CS, Curado MP, Dahlawi SMA, Damiani G, Darwish AH, Daryani A, das Neves J, Demeke FM, Demis AB, Demissie BW, Demoz GT, Denova-Gutierrez E, Derakhshani A, Deribe KS, Desai R, Desalegn BB, Desta M, Dey S, Dharmaratne SD, Dhimal M, Diaz D, Dinberu MTT, Djalalinia S, Doku DT, Drake TM, Dubey M, Dubljanin E, Duken EE, Ebrahimi H, Effiong A, Eftekhari A, El Sayed I, Zaki MES, El-Jaafary SI, El-Khatib Z, Elemineh DA, Elkout H, Ellenbogen RG, Elsharkawy A, Emamian MH, Endalew DA, Endries AY, Eshrati B, Fadhil I, Fallah Omrani V, Faramarzi M, Farhangi MA, Farioli A, Farzadfar F, Fentahun N, Fernandes E, Feyissa GT, Filip I, Fischer F, Fisher JL, Force LM, Foroutan M, Freitas M, Fukumoto T, Futran ND, Gallus S, Gankpe FG, Gayesa RT, Gebrehiwot TT, Gebremeskel GG, Gedefaw GA, Gelaw BK, Geta B, Getachew S, Gezae KE, Ghafourifard M, Ghajar A, Ghashghaee A, Gholamian A, Gill PS, Ginindza TTG, Girmay A, Gizaw M, Gomez RS, Gopalani SV, Gorini G, Goulart BNG, Grada A, Ribeiro Guerra M, Guimaraes ALS, Gupta PC, Gupta R, Hadkhale K, Haj-Mirzaian A, Haj-Mirzaian A, Hamadeh RR, Hamidi S, Hanfore LK, Haro JM, Hasankhani M, Hasanzadeh A, Hassen HY, Hay RJ, Hay SI, Henok A, Henry NJ, Herteliu C, Hidru HD, Hoang CL, Hole MK, Hoogar P, Horita N, Hosgood HD, Hosseini M, Hosseinzadeh M, Hostiuc M, Hostiuc S, Househ M, Hussen MM, Ileanu B, Ilic MD, Innos K, Irvani SSN, Iseh KR, Islam SMS, Islami F, Jafari Balalami N, Jafarinia M, Jahangiry L, Jahani MA, Jahanmehr N, Jakovljevic M, James SL, Javanbakht M, Jayaraman S, Jee SH, Jenabi E, Jha RP, Jonas JB, Jonnagaddala J, Joo T, Jungari SB, Jurisson M, Kabir A, Kamangar F, Karch A, Karimi N, Karimian A, Kasaeian A, Kasahun GG, Kassa B, Kassa TD, Kassaw MW, Kaul A, Keiyoro PN, Kelbore AG, Kerbo AA, Khader YS, Khalilarjmandi M, Khan EA, Khan G, Khang YH, Khatab K, Khater A, Khayamzadeh M, Khazaee-Pool M, Khazaei S, Khoja AT, Khosravi MH, Khubchandani J, Kianipour N, Kim D, Kim YJ, Kisa A, Kisa S, Kissimova-Skarbek K, Komaki H, Koyanagi A, Krohn KJ, Bicer BK, Kugbey N, Kumar V, Kuupiel D, La Vecchia C, Lad DP, Lake EA, Lakew AM, Lal DK, Lami FH, Lan Q, Lasrado S, Lauriola P, Lazarus JV, Leigh J, Leshargie CT, Liao Y, Limenih MA, Listl S, Lopez AD, Lopukhov PD, Lunevicius R, Madadin M, Magdeldin S, El Razek HMA, Majeed A, Maleki A, Malekzadeh R, Manafi A, Manafi N, Manamo WA, Mansourian M, Mansournia MA, Mantovani LG, Maroufizadeh S, Martini SMS, Mashamba-Thompson TP, Massenburg BB, Maswabi MT, Mathur MR, McAlinden C, McKee M, Meheretu HAA, Mehrotra R, Mehta V, Meier T, Melaku YA, Meles GG, Meles HG, Melese A, Melku M, Memiah PTN, Mendoza W, Menezes RG, Merat S, Meretoja TJ, Mestrovic T, Miazgowski B, Miazgowski T, Mihretie KMM, Miller TR, Mills EJ, Mir SM, Mirzaei H, Mirzaei HR, Mishra R, Moazen B, Mohammad DK, Mohammad KA, Mohammad Y, Darwesh AM, Mohammadbeigi A, Mohammadi H, Mohammadi M, Mohammadian M, Mohammadian-Hafshejani A, Mohammadoo-Khorasani M, Mohammadpourhodki R, Mohammed AS, Mohammed JA, Mohammed S, Mohebi F, Mokdad AH, Monasta L, Moodley Y, Moosazadeh M, Moossavi M, Moradi G, Moradi-Joo M, Moradi-Lakeh M, Moradpour F, Morawska L, Morgado-da-Costa J, Morisaki N, Morrison SD, Mosapour A, Mousavi SM, Muche AA, Muhammed OSS, Musa J, Nabhan AF, Naderi M, Nagarajan AJ, Nagel G, Nahvijou A, Naik G, Najafi F, Naldi L, Nam HS, Nasiri N, Nazari J, Negoi I, Neupane S, Newcomb PA, Nggada HA, Ngunjiri JW, Nguyen CT, Nikniaz L, Ningrum DNA, Nirayo YL, Nixon MR, Nnaji CA, Nojomi M, Nosratnejad S, Shiadeh MN, Obsa MS, Ofori-Asenso R, Ogbo FA, Oh IH, Olagunju AT, Olagunju TO, Oluwasanu MM, Omonisi AE, Onwujekwe OE, Oommen AM, Oren E, Ortega-Altamirano DDV, Ota E, Otstavnov SS, Owolabi MO, P A M, Padubidri JR, Pakhale S, Pakpour AH, Pana A, Park EK, Parsian H, Pashaei T, Patel S, Patil ST, Pennini A, Pereira DM, Piccinelli C, Pillay JD, Pirestani M, Pishgar F, Postma MJ, Pourjafar H, Pourmalek F, Pourshams A, Prakash S, Prasad N, Qorbani M, Rabiee M, Rabiee N, Radfar A, Rafiei A, Rahim F, Rahimi M, Rahman MA, Rajati F, Rana SM, Raoofi S, Rath GK, Rawaf DL, Rawaf S, Reiner RC, Renzaho AMN, Rezaei N, Rezapour A, Ribeiro AI, Ribeiro D, Ronfani L, Roro EM, Roshandel G, Rostami A, Saad RS, Sabbagh P, Sabour S, Saddik B, Safiri S, Sahebkar A, Salahshoor MR, Salehi F, Salem H, Salem MR, Salimzadeh H, Salomon JA, Samy AM, Sanabria J, Santric Milicevic MM, Sartorius B, Sarveazad A, Sathian B, Satpathy M, Savic M, Sawhney M, Sayyah M, Schneider IJC, Schottker B, Sekerija M, Sepanlou SG, Sepehrimanesh M, Seyedmousavi S, Shaahmadi F, Shabaninejad H, Shahbaz M, Shaikh MA, Shamshirian A, Shamsizadeh M, Sharafi H, Sharafi Z, Sharif M, Sharifi A, Sharifi H, Sharma R, Sheikh A, Shirkoohi R, Shukla SR, Si S, Siabani S, Silva DAS, Silveira DGA, Singh A, Singh JA, Sisay S, Sitas F, Sobngwi E, Soofi M, Soriano JB, Stathopoulou V, Sufiyan MB, Tabares-Seisdedos R, Tabuchi T, Takahashi K, Tamtaji OR, Tarawneh MR, Tassew SG, Taymoori P, Tehrani-Banihashemi A, Temsah MH, Temsah O, Tesfay BE, Tesfay FH, Teshale MY, Tessema GA, Thapa S, Tlaye KG, Topor-Madry R, Tovani-Palone MR, Traini E, Tran BX, Tran KB, Tsadik AG, Ullah I, Uthman OA, Vacante M, Vaezi M, Varona Perez P, Veisani Y, Vidale S, Violante FS, Vlassov V, Vollset SE, Vos T, Vosoughi K, Vu GT, Vujcic IS, Wabinga H, Wachamo TM, Wagnew FS, Waheed Y, Weldegebreal F, Weldesamuel GT, Wijeratne T, Wondafrash DZ, Wonde TE, Wondmieneh AB, Workie HM, Yadav R, Yadegar A, Yadollahpour A, Yaseri M, Yazdi-Feyzabadi V, Yeshaneh A, Yimam MA, Yimer EM, Yisma E, Yonemoto N, Younis MZ, Yousefi B, Yousefifard M, Yu C, Zabeh E, Zadnik V, Moghadam TZ, Zaidi Z, Zamani M, Zandian H, Zangeneh A, Zaki L, Zendehdel K, Zenebe ZM, Zewale TA, Ziapour A, Zodpey S, Murray CJL. Global, Regional, and National Cancer Incidence, Mortality, Years of Life Lost, Years Lived With Disability, and Disability-Adjusted Life-Years for 29 Cancer Groups, 1990 to 2017: A Systematic Analysis for the Global Burden of Disease Study. JAMA Oncol. 2019 Dec 1;5(12):1749-1768. doi: 10.1001/jamaoncol.2019.2996. PMID 31560378
- [Result] Planchard D, Popat S, Kerr K, Novello S, Smit EF, Faivre-Finn C, Mok TS, Reck M, Van Schil PE, Hellmann MD, Peters S; ESMO Guidelines Committee. Metastatic non-small cell lung cancer: ESMO Clinical Practice Guidelines for diagnosis, treatment and follow-up. Ann Oncol. 2018 Oct 1;29(Suppl 4):iv192-iv237. doi: 10.1093/annonc/mdy275. No abstract available. PMID 30285222
- [Result] Duma N, Santana-Davila R, Molina JR. Non-Small Cell Lung Cancer: Epidemiology, Screening, Diagnosis, and Treatment. Mayo Clin Proc. 2019 Aug;94(8):1623-1640. doi: 10.1016/j.mayocp.2019.01.013. PMID 31378236
- [Result] Herbst RS, Giaccone G, de Marinis F, Reinmuth N, Vergnenegre A, Barrios CH, Morise M, Felip E, Andric Z, Geater S, Ozguroglu M, Zou W, Sandler A, Enquist I, Komatsubara K, Deng Y, Kuriki H, Wen X, McCleland M, Mocci S, Jassem J, Spigel DR. Atezolizumab for First-Line Treatment of PD-L1-Selected Patients with NSCLC. N Engl J Med. 2020 Oct 1;383(14):1328-1339. doi: 10.1056/NEJMoa1917346. PMID 32997907
- [Result] Mok TSK, Wu YL, Kudaba I, Kowalski DM, Cho BC, Turna HZ, Castro G Jr, Srimuninnimit V, Laktionov KK, Bondarenko I, Kubota K, Lubiniecki GM, Zhang J, Kush D, Lopes G; KEYNOTE-042 Investigators. Pembrolizumab versus chemotherapy for previously untreated, PD-L1-expressing, locally advanced or metastatic non-small-cell lung cancer (KEYNOTE-042): a randomised, open-label, controlled, phase 3 trial. Lancet. 2019 May 4;393(10183):1819-1830. doi: 10.1016/S0140-6736(18)32409-7. Epub 2019 Apr 4. PMID 30955977
- [Result] Wang J, Fei K, Jing H, Wu Z, Wu W, Zhou S, Ni H, Chen B, Xiong Y, Liu Y, Peng B, Yu D, Jiang H, Liu J. Durable blockade of PD-1 signaling links preclinical efficacy of sintilimab to its clinical benefit. MAbs. 2019 Nov-Dec;11(8):1443-1451. doi: 10.1080/19420862.2019.1654303. Epub 2019 Sep 3. PMID 31402780
- [Result] Yang Y, Wang Z, Fang J, Yu Q, Han B, Cang S, Chen G, Mei X, Yang Z, Ma R, Bi M, Ren X, Zhou J, Li B, Song Y, Feng J, Li J, He Z, Zhou R, Li W, Lu Y, Wang Y, Wang L, Yang N, Zhang Y, Yu Z, Zhao Y, Xie C, Cheng Y, Zhou H, Wang S, Zhu D, Zhang W, Zhang L. Efficacy and Safety of Sintilimab Plus Pemetrexed and Platinum as First-Line Treatment for Locally Advanced or Metastatic Nonsquamous NSCLC: a Randomized, Double-Blind, Phase 3 Study (Oncology pRogram by InnovENT anti-PD-1-11). J Thorac Oncol. 2020 Oct;15(10):1636-1646. doi: 10.1016/j.jtho.2020.07.014. Epub 2020 Aug 8. PMID 32781263
- [Result] Yang Y, Sun J, Wang Z, Fang J, Yu Q, Han B, Cang S, Chen G, Mei X, Yang Z, Ma R, Bi M, Ren X, Zhou J, Li B, Song Y, Feng J, Li J, He Z, Zhou R, Li W, Lu Y, Zhou H, Wang S, Sun L, Puig O, Mancao C, Peng B, Fang W, Xu W, Zhang L. Updated Overall Survival Data and Predictive Biomarkers of Sintilimab Plus Pemetrexed and Platinum as First-Line Treatment for Locally Advanced or Metastatic Nonsquamous NSCLC in the Phase 3 ORIENT-11 Study. J Thorac Oncol. 2021 Dec;16(12):2109-2120. doi: 10.1016/j.jtho.2021.07.015. Epub 2021 Aug 3. PMID 34358724
- [Result] Hegde PS, Wallin JJ, Mancao C. Predictive markers of anti-VEGF and emerging role of angiogenesis inhibitors as immunotherapeutics. Semin Cancer Biol. 2018 Oct;52(Pt 2):117-124. doi: 10.1016/j.semcancer.2017.12.002. Epub 2017 Dec 8. PMID 29229461
- [Result] Chen DS, Hurwitz H. Combinations of Bevacizumab With Cancer Immunotherapy. Cancer J. 2018 Jul/Aug;24(4):193-204. doi: 10.1097/PPO.0000000000000327. PMID 30119083
- See also: JAMA Oncol,2019 Dec 1;5(12):1749-1768. doi: 10.1001/jamaoncol.2019.2996 — https://pubmed.ncbi.nlm.nih.gov/31560378/
- See also: Ann Oncol,2018 Oct 1;29(Suppl 4):iv192-iv237. doi: 10.1093/annonc/mdy275 — https://pubmed.ncbi.nlm.nih.gov/30285222/
- See also: Mayo Clin Proc,2019 Aug;94(8):1623-1640. doi: 10.1016/j.mayocp.2019.01.013. — https://pubmed.ncbi.nlm.nih.gov/31378236/
- See also: N Engl J Med,2020 Oct 1;383(14):1328-1339. doi: 10.1056/NEJMoa1917346. — https://pubmed.ncbi.nlm.nih.gov/32997907/
- See also: Lancet,2019 May 4;393(10183):1819-1830. doi: 10.1016/S0140-6736(18)32409-7. Epub 2019 Apr 4. — https://pubmed.ncbi.nlm.nih.gov/30955977/
- See also: MAbs,2019 Nov-Dec;11(8):1443-1451. — https://pubmed.ncbi.nlm.nih.gov/31402780/
- See also: J Thorac Oncol,2020 Oct;15(10):1636-1646. — https://pubmed.ncbi.nlm.nih.gov/32781263/
- See also: J Thorac Oncol . 2021 Dec;16(12):2109-2120. doi: 10.1016/j.jtho.2021.07.015. Epub 2021 Aug 3. — https://pubmed.ncbi.nlm.nih.gov/34358724/
- See also: Semin Cancer Biol . 2018 Oct;52(Pt 2):117-124. doi: 10.1016/j.semcancer.2017.12.002. Epub 2017 Dec 8. — https://pubmed.ncbi.nlm.nih.gov/29229461/
- See also: Cancer J . 2018 Jul/Aug;24(4):193-204. — https://pubmed.ncbi.nlm.nih.gov/30119083/
- Available data/document: Clinical Study Report: [ PMID ]31560378 — https://pubmed.ncbi.nlm.nih.gov/31560378/
- Available data/document: Clinical Study Report: PMID:30285222 — https://pubmed.ncbi.nlm.nih.gov/30285222/
- Available data/document: Clinical Study Report: PMID:31378236 — https://pubmed.ncbi.nlm.nih.gov/31378236/
- Available data/document: Clinical Study Report: PMID:32997907 — https://pubmed.ncbi.nlm.nih.gov/32997907/
- Available data/document: Clinical Study Report: PMID:30955977 — https://pubmed.ncbi.nlm.nih.gov/30955977/
- Available data/document: Clinical Study Report: PMID:31402780 — https://pubmed.ncbi.nlm.nih.gov/31402780/
- Available data/document: Clinical Study Report: PMID:32781263 — https://pubmed.ncbi.nlm.nih.gov/32781263/
- Available data/document: Clinical Study Report: PMID: 34358724 — https://pubmed.ncbi.nlm.nih.gov/34358724/
- Available data/document: Clinical Study Report: PMID: 29229461 — https://pubmed.ncbi.nlm.nih.gov/29229461/
- Available data/document: Clinical Study Report: PMID: 30119083 — https://pubmed.ncbi.nlm.nih.gov/30119083/